CLINICAL TRIAL: NCT04438590
Title: The Use of Kelulut Honey for Carbohydrate-Loading in the Preoperative Period for Patients Undergoing Abdominal Surgery Involving the Digestive System as Part of Enhanced Recovery After Surgery as Opposed to VALENS® Carborie®Load
Brief Title: Kelulut Honey as an Alternate Source of Carbo-Loading in Abdominal Surgery Involving the Digestive System
Acronym: Kel-Load
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, B. Karthik Krishnan, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USMKK
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Insulin Resistance; ERAS
Keywords: carbohydrate loading; honey; insulin resistance; stingless bee; ERAS
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kelulut Honey (Experimental): Medical Grade Kelulut Honey which will be in 2 doses.
  The first would be diluted to 800 ml of water, and the second dose in 400ml of water.
  Interventions: Dietary Supplement: Kelulut Honey
- Carborie (Active Comparator): Carborie Load which will be 100g of carbohydrate in 800 ML of water and 50g of carbohydrate in 400ml of water.
  Interventions: Dietary Supplement: Carborie

INTERVENTIONS:
Dietary Supplement: Kelulut Honey — The Substance being tested to be used as an alternative
  Arms: Kelulut Honey
Dietary Supplement: Carborie — The commercially available substance
  Arms: Carborie

SUMMARY:
The study aims to identify if Kelulut Honey can be a potential alternative for the use of preoperative carboloading instead of the commercially available product, Carborie.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery is a well-established, evidence based multimodal, multidisciplinary approach to the care of the surgical patient. The aim of the program, as per its nomenclature, is to establish a set of protocol to subject the surgical patient to in order to facilitate recovery, attenuate the metabolic responses from surgery, reduce complications and ultimately reduce length of stay as well as establish return of physiological function of the patient in an accelerated fashion.

As mentioned, given that ERAS involves a multimodal, multidisciplinary approach, there are many aspects and guidelines as to the implementation of ERAS. One particular modern care change is conversion of the surgical dogma of overnight fasting to carbo-loading; whereby the patient is subjected to consume a carbohydrate rich drink the evening prior to surgery, and 2 hours prior to induction with anaesthesia. The doctrine of overnight fasting or rather 6-8 hours of fasting has long been the core principal for many anaesthesiologists and surgeons, given the rationale that this would reduce gastric acidity and volume, thereby reducing the risk of vomiting and gastric content aspiration. However, modern guidelines have shown that there are no evidence that shortened fast of 2-3 of oral fluids increase the risk of aspiration, regurgitation or increase morbidity as compared with fasting after midnight.

The problem with fasting, is that it increases insulin resistance. In line with acute-phase response, and loss of lean body mass, this will attenuate the affects of prolonged fasting. So, in an insulin resistant state, cell glucose uptake is reduced, and therefore glycogen formation reduces, which means, the liver and muscle glycogen storage are depleted. Hyperglycaemia ensues, due to the enhanced endogenous glucose production. Glucose control needs to be adequate to avoid risk of surgical complication and mortality.

The benefits of carbo-loading is well documented and the evidence is overwhelming. The evidence shows that oral ingestion of 50g of Carbohydrate has been shown to release Insulin similar to that of a mixed meal. The current guideline advocates 100g of carbohydrate consumed the evening prior to surgery and another 50g 2 hours before surgery. The first dose is consumed with 800 mL of water, and the subsequent dose with 400mL.

Kelulut honey is a natural product, which contains sugar in the form of fructose and glucose produced by bees (Meliponini Sp). They have a rapid onset, as they are freely absorbed into the blood stream without requiring digestion. Honey also has a proven role in facilitating wound healing, and as an anti-inflammatory, and antibacterial agent. The aim of this study is to evaluate the use of honey as an alternative to maltodextrin extract for carbo-loading in patients undergoing elective gastrointestinal surgery (Upper GI and Lower GI) and its effects.

ELIGIBILITY:
Inclusion Criteria

* Adult (Age ≥ 18)
* Elective Surgery with Intraabdominal Involvement

Exclusion Criteria

* Known Diabetics
* Fasting Glucose Level > 7 mmol/L
* ASA > 3
* On Steroid Treatment
* Recent Infection Past 3 Months
* Preoperative Unintentional Weight Loss >10% of usual body weight within 6 months
* Emergency Surgery
* Minor (Age < 18)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Kelulut Honey Improves Insulin Resistance when used as carbo-loading preoperatively | 48 Hours
  • To compare blood sugar levels between patients receiving Kelulut Honey and Carborie pre, intra, and post operatively.
Kelulut Honey would be completely cleared within 2 hours after consumption when used for carbo-loading preoperatively. | 2 hours
  • To compare Residual Gastric Volume between patients receiving Kelulut Honey and Carborie preoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liz Goldenberg., Fasting versus Carb-Loading: What's the Evidence for Your Enhanced Recovery after Bariatric Surgery Program?, Bariatric Times. 2018;15(11):28-29
- [Result] Yagci G, Can MF, Ozturk E, Dag B, Ozgurtas T, Cosar A, Tufan T. Effects of preoperative carbohydrate loading on glucose metabolism and gastric contents in patients undergoing moderate surgery: a randomized, controlled trial. Nutrition. 2008 Mar;24(3):212-6. doi: 10.1016/j.nut.2007.11.003. Epub 2007 Dec 21. PMID 18096368
- [Result] Scott MJ, Fawcett WJ. Oral carbohydrate preload drink for major surgery - the first steps from famine to feast. Anaesthesia. 2014 Dec;69(12):1308-13. doi: 10.1111/anae.12921. Epub 2014 Oct 23. No abstract available. PMID 25346490
- [Result] Nakamura M, Uchida K, Akahane M, Watanabe Y, Ohtomo K, Yamada Y. The effects on gastric emptying and carbohydrate loading of an oral nutritional supplement and an oral rehydration solution: a crossover study with magnetic resonance imaging. Anesth Analg. 2014 Jun;118(6):1268-73. doi: 10.1213/ANE.0b013e3182a9956f. PMID 24384864
- [Result] Mustafa MZ, Yaacob NS, Sulaiman SA. Reinventing the Honey Industry: Opportunities of the Stingless Bee. Malays J Med Sci. 2018 Jul;25(4):1-5. doi: 10.21315/mjms2018.25.4.1. Epub 2018 Aug 30. PMID 30914843
- [Result] Maitra S, Kirtania J, Pal S, Bhattacharjee S, Layek A, Ray S. Intraoperative blood glucose levels in nondiabetic patients undergoing elective major surgery under general anaesthesia receiving different crystalloid solutions for maintenance fluid. Anesth Essays Res. 2013 May-Aug;7(2):183-8. doi: 10.4103/0259-1162.118953. PMID 25885830
- [Result] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Result] Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, von Meyenfeldt MF, Fearon KC, Revhaug A, Norderval S, Ljungqvist O, Lobo DN, Dejong CH; Enhanced Recovery After Surgery (ERAS) Group. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Arch Surg. 2009 Oct;144(10):961-9. doi: 10.1001/archsurg.2009.170. PMID 19841366
- [Result] Kratzing C. Pre-operative nutrition and carbohydrate loading. Proc Nutr Soc. 2011 Aug;70(3):311-5. doi: 10.1017/S0029665111000450. PMID 21781358
- [Result] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Result] Gianotti L, Biffi R, Sandini M, Marrelli D, Vignali A, Caccialanza R, Vigano J, Sabbatini A, Di Mare G, Alessiani M, Antomarchi F, Valsecchi MG, Bernasconi DP. Preoperative Oral Carbohydrate Load Versus Placebo in Major Elective Abdominal Surgery (PROCY): A Randomized, Placebo-controlled, Multicenter, Phase III Trial. Ann Surg. 2018 Apr;267(4):623-630. doi: 10.1097/SLA.0000000000002325. PMID 28582271
- [Result] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- [Result] Zulkhairi Amin FA, Sabri S, Mohammad SM, Ismail M, Chan KW, Ismail N, Norhaizan ME, Zawawi N. Therapeutic Properties of Stingless Bee Honey in Comparison with European Bee Honey. Adv Pharmacol Sci. 2018 Dec 26;2018:6179596. doi: 10.1155/2018/6179596. eCollection 2018. PMID 30687402
- [Result] Sudiyatmo, et al., Effects of Preoperative Honey Drink on Gastric Content, Perioperative Discomfort and Insulin Resistance in Patients Undergoing Open Colorectal Surgery a Randomized, Controlled Trial. British Journal of Medicine & Medical Research, 14(7): 1-8, 2016.
- [Result] Abdul JA, et al., Surgical Services In Malaysian Hospitals. National Healthcare Establishment & Workforce Statistics (NHEWS) 2011, NCRC/HSU/2013.1 C4:47-63, 2013